CLINICAL TRIAL: NCT06179290
Title: A Multi-site, Open-Label, Parallel-Group Study To Evaluate Changes In Tobacco-Related Biomarkers of Exposure and Biomarkers of Potential Harm With Use of Heated Tobacco Products Compared to Combustible Cigarettes in Adult Smokers
Brief Title: Changes in Biomarker of Exposure in Adults Who Smoke Cigarettes Switching From Cigarettes to Heated Tobacco Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altria Client Services LLC (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ALCS-REG-23-07-HT
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use
Keywords: Tobacco; Smoking; Heated tobacco
MeSH Terms: conditions — Tobacco Use; Smoking | interventions — Menthol

STUDY DESIGN:
Intervention Model Description: This is a multi-site, open-label, two-group (menthol and non-menthol), six-arm (HTP, Continue Smoking, and Smoking Abstinence arms within each group) randomized, clinical study to evaluate changes in BoEs in adult smokers who remain smoking, switch to the Ploom HTP, or abstain from smoking, for 60 days (5 days in clinic followed by 55-day ambulatory phase). This study follows the recommendations of the FDA's final Premarket Tobacco Product Application guidance (FDA, 2023).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Study Product A: Ploom HTP Menthol HTS; MX3 (681) (Experimental): Subjects in A arm (Group 1 Menthol) will be required to smoke Ploom HTP Menthol HTS; MX3 (681) study product at least 5 times per day ad libitum from 07:00 through 23:00. There will be 60 subjects assigned to this arm with a randomization ratio of 2.
  Interventions: Other: Ploom HTP Menthol HTS; MX3 (681)
- Study Product B: Continue Smoking (menthol) (No Intervention): Subjects in B arm (Group 1 Menthol) will continue to smoke their menthol UBCC ad libitum from 07:00 through 23:00. There will be 60 subjects assigned to this arm with a randomization ratio of 2.
- Study Product C: Smoking Abstinence (menthol) (Active Comparator): Subjects in C arm (Group 1 Menthol) will remain abstinent from cigarette smoking for the duration of the study during both the confinement and ambulatory phases. There will be 30 subjects assigned to this arm with a randomization ratio of 1.
  Interventions: Other: Smoking Abstinence (menthol)
- Study Product D: Ploom HTP Tobacco HTS; R8 (120) (Experimental): Subjects in D arm (Group 2 Non-menthol) will be required to smoke Ploom HTP Tobacco HTS; R8 (120) study product at least 5 times per day ad libitum from 07:00 through 23:00. There will be 60 subjects assigned to this arm with a randomization ratio of 2.
  Interventions: Other: Ploom HTP Tobacco HTS; R8 (120)
- Study Product E: Continue Smoking (non-menthol) (No Intervention): Subjects in E arm (Group 2 Non-menthol) will continue to smoke their non-menthol UBCC ad libitum from 07:00 through 23:00. There will be 60 subjects assigned to this arm with a randomization ratio of 2.
- Study Product F: Smoking Abstinence (non-menthol) (Active Comparator): Subjects in F arm (Group 2 Non-menthol) will remain abstinent from cigarette smoking for the duration of the study during both the confinement and ambulatory phases. There will be 30 subjects assigned to this arm with a randomization ratio of 1.
  Interventions: Other: Smoking Abstinence (non-menthol)

INTERVENTIONS:
Other: Ploom HTP Menthol HTS; MX3 (681) — Menthol heated tobacco product
  Arms: Study Product A: Ploom HTP Menthol HTS; MX3 (681)
Other: Ploom HTP Tobacco HTS; R8 (120) — Non-menthol heated tobacco product
  Arms: Study Product D: Ploom HTP Tobacco HTS; R8 (120)
Other: Smoking Abstinence (menthol) — No smoking or other tobacco product use for duration of the study, menthol group comparator
  Arms: Study Product C: Smoking Abstinence (menthol)
Other: Smoking Abstinence (non-menthol) — No smoking or other tobacco product use for duration of the study, non-menthol group comparator
  Arms: Study Product F: Smoking Abstinence (non-menthol)

SUMMARY:
The purpose of the study is to evaluate changes in biomarkers of exposure (BoE) to harmful and potentially harmful constituents (HPHCs) in adult smokers who completely switch to Ploom heated tobacco products (HTPs) compared to those who continue to smoke usual brand combustible cigarettes (UBCC).

DETAILED DESCRIPTION:
This is a multi-site, open-label, two-group (menthol and non-menthol), six-arm (HTP, Continue Smoking, and Smoking Abstinence arms within each group) randomized, clinical study to evaluate changes in BoEs in adult smokers who remain smoking, switch to the Ploom HTP, or abstain from smoking, for 60 days (5 days in clinic followed by a 55-day ambulatory phase). Target enrollment is 300 male and female adult smokers between the ages of 22 and 65 in overall good health.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary consent to participate in this study documented on the signed ICF.
2. Score 5 or higher (moderate dependence or higher) on the FTCD.
3. Healthy adult males and females ≥ 22 and ≤ 65 years of age, inclusive, at Screening.
4. Smoking history (self-reported at screening) of an average of at least 10 but no more than 30 factory-manufactured combustible cigarettes (either menthol or non-menthol) daily for at least 12 months prior to screening. Brief periods (ie, up to 7 consecutive days) of non-smoking during the 3 months prior to screening (eg, due to illness or participation in a study where smoking was prohibited) will be permitted.
5. Screening and first check-in blood pressure ≤ 150/90 mmHg measured after being seated for at least 10 minutes. Two rechecks may be performed at the Principal Investigator's discretion.
6. Positive urine cotinine (≥ 500 ng/mL) at screening.
7. Exhaled carbon monoxide (eCO) ≥ 10 ppm at screening.
8. Post-bronchodilator forced expired volume in 1 second (FEV1) : forced vital capacity (FVC) ratio > 0.7 and FEV1 > 80% of predicted at screening.
9. Negative pregnancy test at Screening and first check-in (Day -2) for all female subjects.
10. Female subjects who are heterosexually active and of childbearing potential (eg, neither surgically sterile at least 6 months prior to first check-in nor postmenopausal with amenorrhea for at least 12 months prior to first check-in with follicle-stimulating hormone [FSH] levels consistent with postmenopausal status) must have been using one of the following forms of contraception for the time period indicated and agree to continue using it through completion of the study:

    * hormonal (eg, oral, vaginal ring, transdermal patch, implant, injection) consistently for at least 3 months prior to first check-in, when used in combination with male condoms with spermicide (use of NuvaRing® is at the Principal Investigator's discretion)
    * double barrier (eg, condom with spermicide or diaphragm with spermicide) consistently for at least 2 weeks prior to first check-in
    * intrauterine device or system (utilize Principal Investigator discretion regarding use of hormonal or nonhormonal devices) for at least 3 months prior to first check-in
    * exclusive partner who is clinically sterile (ie, documented infertility or surgical sterilization; see below for additional information on sterility) or has been vasectomized for at least 6 months (inclusive) prior to first check-in Note: Sexual abstinence, defined as refraining from intercourse, is allowed when this is in line with the preferred and usual lifestyle of the subject. Female subjects of childbearing potential who are not currently engaging in heterosexual intercourse must agree to use one of the above methods of birth control through completion of study, in the event that they have heterosexual intercourse during the course of the study.
11. Female subjects who are of nonchildbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to first check-in:

    * Hysteroscopic sterilization (including Essure® or similar nonsurgical sterilization procedures);
    * bilateral tubal ligation or bilateral salpingectomy;
    * hysterectomy;
    * bilateral oophorectomy Or be postmenopausal with amenorrhea for at least 12 months prior to first check-in and have FSH levels consistent with postmenopausal status.
12. Willing to comply with the requirements of the study.
13. Willing to use Ploom HTP after the Product Trial at first check-in.
14. Willing and able to abstain from cigarettes from Day 1 through the end of the study (EOS) on Day 60 (±3 days) if they are randomized to a Smoking Abstinence arm.

Exclusion Criteria:

1. Use of any type of tobacco- or nicotine-containing products other than manufactured cigarettes (eg, e-vapor products, roll-your-own cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) in the 7 days prior to first check-in.
2. Self-reported puffers (ie, adult smokers who draw smoke from the cigarette into the mouth and throat but do not inhale).
3. Planning to quit smoking in the next three months (at screening).
4. History or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, existing respiratory diseases, immunologic, psychiatric, lymphatic, or cardiovascular disease, or any other condition that, in the opinion of the Principal Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
5. Clinically significant abnormal findings on the vital signs, physical examination, medical history, ECG, or clinical laboratory results, in the opinion of the Principal Investigator.
6. Positive test for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus at screening.
7. History or presence of any type of malignant tumors.
8. Current evidence or any history of congestive heart failure.
9. Diabetes mellitus (fasting glucose ≥126 mg/L [7 mmol/L]) that is not controlled by diet/exercise alone, in the opinion of the Principal Investigator.
10. An acute illness (eg, upper respiratory infection, viral infection) requiring treatment with prescribed medicines within 2 weeks prior to first check-in.
11. Any planned surgery from the time of screening through EOS.
12. History of drug or alcohol abuse within 24 months prior to first check-in.
13. Fever (ie, body temperature >100.5°F) at screening or first check-in. One re-check may be performed at the Principal Investigator's discretion.
14. Body mass index greater than 40.0 kg/m2 or less than 18.0 kg/m2 at screening.
15. Systolic blood pressure >150 mmHg and/or diastolic blood pressure > 90 mmHg at screening or first check-in, measured after being seated for at least 10 minutes. Two re-checks may be performed at the Principal Investigator's discretion.
16. Estimated creatinine clearance (by Cockcroft-Gault equation) < 80 mL/minute at screening.
17. Serum alanine aminotransferase ≥1.5 times the upper limit of normal and/or aspartate aminotransferase ≥1.5 times the upper limit of normal at screening.
18. Positive screen for alcohol (urine/breath) or any of the following drugs of abuse (urine/saliva), regardless of the reason of use: amphetamines, methamphetamines, opiates, cannabinoids, or cocaine at screening or first check-in.
19. Female subjects who are pregnant (positive serum pregnancy test at screening or urine/serum pregnancy test at first check-in), lactating, or intend to become pregnant from screening through EOS.
20. Use of prescription or over-the-counter bronchodilator medication (eg, inhaled or oral ß-agonists) for treatment of any illnesses and within 12 months prior to first check-in and throughout the study.
21. Use of medications or foods known or are suspected to interact with cytochrome P450 2A6 (including, but not limited to, amiodarone, amlodipine, amobarbital, clofibrate, clotrimazole, desipramine, disulfiram, entacapone, fenofibrate, isoniazid, grapefruit, ketoconazole, letrozole, methimazole, methoxsalen, metyrapone, miconazole, modafinil, orphenadrine, pentobarbital, phenobarbital, pilocarpine, primidone, propoxyphene, quinidine, rifampicin, rifampin, secobarbital, selegiline, sulconazole, tioconazole, tranylcypromine) within 14 days or 5 half-lives of the drug, whichever is longer, prior to first check-in or during the study.
22. Use of antibiotic treatment within 2 weeks prior to first check-in.
23. Plasma donation within 7 days prior to first check-in.
24. Donation of blood or blood products (with the exception of plasma as noted above), had significant blood loss, or received whole blood or a blood product transfusion within 56 days prior to first check-in.
25. Participation in a previous clinical study for an investigational drug, device, biologic, or a tobacco product within 30 days prior to first check-in.
26. Subject or a first-degree relative (ie, parent, sibling, child, spouse/partner) is a current or former employee of the tobacco industry or a named party or class representative in litigation with any tobacco company.
27. Subject or a first-degree relative (ie, parent, sibling, child, spouse/partner) is a current employee of the study site.
28. Have been diagnosed with major depressive disorder or have a history of suicide attempt.
29. Have pre-bronchodilator to post-bronchodilator FEV1 increases of greater than or equal to 12% or grade "C" or worse per ATS/ERS 2019 standards.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 921 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) | Baseline through Day 5
  Total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) in urine
Total N-nitrosonornicotine (NNN) | Baseline through Day 5
  Total N-nitrosonornicotine (NNN) in urine
2-hydroxybutenylmercapturic acid (2-MHBMA) | Baseline through Day 5
  2-hydroxybutenylmercapturic acid (2-MHBMA) in urine
3-hydroxypropylmercapturic acid (3-HPMA) | Baseline through Day 5
  3-hydroxypropylmercapturic acid (3-HPMA) in urine
S-phenyl mercapturic acid (SPMA) | Baseline through Day 5
  S-phenyl mercapturic acid (SPMA) in urine
2-Hydroxyethyl mercapturic acid (HEMA) | Baseline through Day 5
  2-Hydroxyethyl mercapturic acid (HEMA) in urine
1-aminonaphthalene (1-AN) | Baseline through Day 5
  1-aminonaphthalene (1-AN) in urine
2-aminonaphthalene (2-AN) | Baseline through Day 5
  2-aminonaphthalene (2-AN) in urine
2-cyanoethyl-mercapturic acid (CEMA) | Baseline to Day 5
  2-cyanoethyl-mercapturic acid (CEMA) in urine
3-hydroxybenzo[a]pyrene (3-OH-B[a]P) | Baseline through Day 5
  3-hydroxybenzo[a]pyrene (3-OH-B[a]P) in urine
3-hydroxy-1-methylpropylmercapturic acid (HMPMA) | Baseline through Day 5
  3-hydroxy-1-methylpropylmercapturic acid (HMPMA) in urine
4-Aminobiphenyl (4-ABP) | Baseline through Day 5
  4-Aminobiphenyl (4-ABP) in urine
S-benzyl mercapturic acid (SBMA) | Baseline through Day 5
  S-benzyl mercapturic acid (SBMA) in urine
Carboxyhemoglobin (COHb) | Baseline to Day 5
  Carboxyhemoglobin (COHb) in blood

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Woodland Research Northwest, Rogers, Arkansas
  - Dr. Vince Clinical Research, LLC, Overland Park, Kansas
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - QPS Bio-Kinetic, Springfield, Missouri
  - Celerion Lincoln, Lincoln, Nebraska
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Spaulding Clinical Research, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: No